CLINICAL TRIAL: NCT03581630
Title: Effects of Mediterranean Diet and Naltrexone/Bupropion Treatment on Body Weight and Metabolic Risk Factors in Obese Breast Cancer Patients After Breast Cancer Treatment
Brief Title: Effects of Mediterranean Diet and Naltrexone/Bupropion Treatment in Obese Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Associate Professor (Department of Family Medicine, Gangnam Severance Hospital,, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3-2017-0097
Record Dates: First submitted 2018-05-15; First posted 2018-07-10 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Obesity; Overweight
MeSH Terms: conditions — Breast Neoplasms; Obesity; Overweight | interventions — Naltrexone; Bupropion; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast cancer subjects-naltrexone/bupropion+Mediterranean Diet (Experimental)
  Interventions: Drug: naltrexone/bupropion; Behavioral: Mediterranean Diet
- Breast cancer subjects-Mediterranean Diet (Experimental)
  Interventions: Behavioral: Mediterranean Diet
- Healthy subjects-naltrexone/bupropion+Mediterranean Diet (Active Comparator)
  Interventions: Drug: naltrexone/bupropion; Behavioral: Mediterranean Diet

INTERVENTIONS:
Drug: naltrexone/bupropion — Naltrexone hydrochloride (HCl) 8 mg/Bupropion hydrochloride (HCl) 90 mg extended release (ER) combination tablets, orally, one tablet, in the morning, daily, for 1 week, followed by Naltrexone HCl 8 mg/Bupropion HCl 90 mg ER combination tablets, orally, one tablet in the morning and one in the evening, daily, for 7 weeks.
  Arms: Breast cancer subjects-naltrexone/bupropion+Mediterranean Diet; Healthy subjects-naltrexone/bupropion+Mediterranean Diet
Behavioral: Mediterranean Diet — Diet instruction and menu samples from the dietitian on following the Mediterranean Diet.

SUMMARY:
Obesity among breast cancer survivors is known to be associated with recurrence and other co-morbidities. However, there have been no studies on weight reduction program combining diet and anti-obesity drug for obese breast cancer survivors. The purpose of this randomized clinical trial is to examine the effects of Mediterranean Diet and naltrexone/bupropion treatment on inflammation and metabolic risk factors in overweight or obese breast cancer patients after breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female, 20 to 65 years of age
* Diagnosed with breast cancer stage Ⅰ-Ⅲ, and have completed cancer treatment including breast surgery and/or adjuvant chemotherapy, radiotherapy, hormonal therapy
* BMI ≥25 kg/m2, or BMI ≥23 kg/m2 with one or more of the metabolic risk factors (waist circumference ≥80 cm, fasting glucose ≥100 mg/dL, BP ≥130/85 mmHg, HDL-cholesterol <50 mg/dL or controlled diabetes, hypertension, dyslipidemia with medications)
* If woman of child bearing potential, agree to use effective contraception throughout the study period and 30 days after discontinuation of study drug
* Able to speak and read Korean
* Able to comply with all required study procedures and schedule
* Willing and able to give written informed consent

Exclusion Criteria:

* Participants with cancer recurrence or metastasis
* Participants with uncontrolled hypertension (systolic blood pressure (SBP) >180 mmHg, or diastolic blood pressure (DBP) >120 mmHg)
* Participants with hepatic disease (aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >3 x institutional upper limit of normal) or renal disease (serum creatinine >2.0 mg/dL)
* Participants with significant cardiovascular disease or stroke
* Participants with history of seizures
* Participants with serious psychiatric illness, including bipolar disorder, schizophrenia, or other psychosis, bulimia, anorexia nervosa, or suicidal ideation
* Participants who are taking medications such as monoamine oxidase (MAO) inhibitors, opioid-containing medications, other naltrexone or bupropion containing medications, and Tamoxifen
* Current smokers or use of nicotine replacement products in the previous 6 months
* Pregnant or breast-feeding women
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-07-22 (Actual)

PRIMARY OUTCOMES:
Change in body weight | baseline, 8 weeks
  body weight (kg)
Change in fat mass | baseline, 8 weeks
  fat mass (kg) measured by bioelectrical impedance analyzer
Change in muscle mass | baseline, 8 weeks
  muscle mass (kg) measured by bioelectrical impedance analyzer
Change in fasting glucose | baseline, 8 weeks
  fasting glucose (mg/dL)
Change in insulin | baseline, 8 weeks
  insulin (mcIU/mL)
Change in triglyceride | baseline, 8 weeks
  triglyceride (mg/dL)
Change in high-density lipoprotein cholesterol (HDL-cholesterol) | baseline, 8 weeks
  HDL-cholesterol (mg/dL)
Change in leukocyte count | baseline, 8 weeks
  leukocyte count (/μL)

CONTACTS AND LOCATIONS:
Overall Officials: ji won Lee, MD. PhD., Principal Investigator — 82-2-2019-3480
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho AR, Choi WJ, Kwon YJ, Lee HS, Ahn SG, Lee JW. Mediterranean Diet and Naltrexone/Bupropion Treatment for Weight Loss in Overweight and Obese Breast Cancer Survivors and Non-Cancer Participants: A Pilot Randomized Controlled Trial. Diabetes Metab Syndr Obes. 2020 Sep 29;13:3325-3335. doi: 10.2147/DMSO.S269237. eCollection 2020. PMID 33061494